CLINICAL TRIAL: NCT01207661
Title: Mesenchymal Stem Cells Transplantation for Articular Cartilage Resurfacing in Patient With Osteoarthritis of Knee Joint
Brief Title: Articular Cartilage Resurfacing With Mesenchymal Stem Cells In Osteoarthritis Of Knee Joint
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Bone-002
Record Dates: First submitted 2010-09-06; First posted 2010-09-23 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2009-04

CONDITIONS: Osteoarthritis
Keywords: Mesenchymal cells; osteoarthritis; intra articular injection
MeSH Terms: conditions — Osteoarthritis | interventions — Carboxylesterase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal Injection (Experimental): Intra Articular injection in Patients with osteoarthritis of knee joint
  Interventions: Biological: Mesenchymal Injection

INTERVENTIONS:
Biological: Mesenchymal Injection — Intra Articular Injection of Mesenchymal cells to the knee joint
  Other Names: Cell Injection

SUMMARY:
Knee osteoarthritis is the most common form of arthritis. Treatments involve high costs in terms of social and economic, are palliative and do not contemplate healing by regenerative therapy. It has been shown recently, that mesenchymal stem cells (MSC) can be expanded in vitro and may regenerate several damaged or injured tissues. In addition its has demonstrated that MSC are able to modulate immune responses and to control inflammation through its action on T lymphocytes. Preliminary studies in animal models, including one carried out in an equine by the investigators research group, confirms feasibility, safety and efficacy evidence proposed treatment protocol.This study is designed to evaluate therapeutic potential and safety of mesenchymal stem cells in improvement of osteoarthritis clinical manifestations.This study is designed to evaluate therapeutic potential and safety of mesenchymal stem cells in improvement of osteoarthritis clinical manifestations.

DETAILED DESCRIPTION:
Mesenchymal stem cells are pluripotent cells that can be obtained from various tissues .They have shown capabilities to differentiate into bone,cartilage,muscle,and adipose tissue, representing a new clinical strategy in regenerative medicine.An increasing number of reports have demonstrated effectiveness of percutaneous intra-articular infusion of MSCs in arthritic disease. In this study we perform a single intra articular injection of cultured mesenchymal stem cells in patients suffering from osteoarthritis, with the aim to assess its clinical safety and efficacy.Patients are assessed for response with MRI, X-Ray examination, WOMAC osteoarthritis index,VAS, and SF36 2,4,8 weeks and 6, and 12 months post infusion.

ELIGIBILITY:
Inclusion Criteria:

* Female patients not pregnant or lactating.
* Patients with a history of corticosteroids or on active therapy, will only be eligible for enrollment if corticosteroid use is suspended for 1 month prior cell therapy
* Marcaine 0.75% و Lidocaine 4% test performed to be assure the exact location of the pain is related to the knee.
* Diagnosis must be based on magnetic resonance imaging.
* Both genders
* Age:18-65 years

Exclusion Criteria:

* Diagnosis of cancer,DM,CNS disorder,thyroid disease or respiratory disease.
* Known allergic reaction to components of study treatment and/or study injection procedure
* Patients infected with hepatitis B,C or HIV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pain relief | 6 months
  evaluation the effect of Mesenchymal stem cell transplantation to decrease the patients pain

SECONDARY OUTCOMES:
Pain relief | 6 months
  decrease the patient pain in VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Mohammad reza Baghban Eslami Nejad, PhD, Study Director — Scientific Board; Mohssen Emadeddin, MD, Principal Investigator — Orthopadic Investigator; Nasser Aghdami, MD,PhD, Principal Investigator — Head of Regeneration center
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Emadedin M, Ghorbani Liastani M, Fazeli R, Mohseni F, Moghadasali R, Mardpour S, Hosseini SE, Niknejadi M, Moeininia F, Aghahossein Fanni A, Baghban Eslaminejhad R, Vosough Dizaji A, Labibzadeh N, Mirazimi Bafghi A, Baharvand H, Aghdami N. Long-Term Follow-up of Intra-articular Injection of Autologous Mesenchymal Stem Cells in Patients with Knee, Ankle, or Hip Osteoarthritis. Arch Iran Med. 2015 Jun;18(6):336-44. PMID 26058927
- See also: Related Info — http://www.royaninstitute.org